CLINICAL TRIAL: NCT05289206
Title: The Effects of the Interchangeability of the Booster Vaccine Against COVID-19 on the Immune Response Among Education and Public Safety Workers With Risk Factors for Severity, in Manaus (Amazonas)
Brief Title: Immune Response of an Interchangeable Booster Vaccine Against COVID-19 Among Individuals With Risk Factors for Severity
Acronym: COVACManaus2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundação de Medicina Tropical Dr. Heitor Vieira Dourado (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Amazonas (FAPEAM) (Unknown); XP Investimentos (Unknown); Universidade do Estado do Amazonas (UEA) (Unknown); Oswaldo Cruz Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CAAE: 51701821.6.0000.0005
Record Dates: First submitted 2021-09-13; First posted 2022-03-21 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Comorbidities and Coexisting Conditions; Healthy
Keywords: Covid19; vaccine; ChAdOx1-S/nCoV-19 [recombinant]
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Experimental, single-arm study in participants with comorbidities, previously immunized with 2 doses of CoronaVac, who will receive a booster vaccine with 1 dose of the Oxford/AstraZeneca vaccine (ChAdOx1-S/nCoV-19 [recombinant]).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention - single arm (Experimental): Oxford/AstraZeneca (ChAdOx1-S/nCoV-19 [recombinant]) - 0.5 mL single dose, intramuscular in deltoid, with an interval of 180 days (+/- 30 days) from the 2nd dose of the initial vaccination schedule with CoronaVac
  Interventions: Other: Vaccine - ChAdOx1-S/nCoV-19 [recombinant]

INTERVENTIONS:
Other: Vaccine - ChAdOx1-S/nCoV-19 [recombinant] — ChAdOx1-S/nCoV-19 [recombinant] - 0.5 mL single dose, intramuscular in deltoid, with an interval of 180 days (+/- 30 days) from the 2nd dose of the initial vaccination schedule with CoronaVac

SUMMARY:
Experimental, single-arm study in participants with comorbidities, previously immunized with 2 doses of CoronaVac, who will receive a booster vaccine with 1 dose of the Oxford/AstraZeneca vaccine.

DETAILED DESCRIPTION:
Intervention: Oxford/AstraZeneca - 0.5 mL single dose, intramuscular in deltoid, with an interval of 180 days (+/- 30 days) from the 2nd dose of the initial vaccination schedule with CoronaVac

Inclusion criteria:

* Have voluntarily participated and be in regular follow-up monitoring by the COVACMANAUS study;
* Have completed the vaccination schedule with 2 doses of CoronaVac, as per the COVACMANAUS study protocol for at least 180 days (+/- 30 days);
* Demonstrate availability to be followed during the follow-up period defined in the study, through visits, telephone contacts or other digital means of communication;
* Accept to participate in this new study for 6 (six) months.

Exclusion criteria

* Confirmed diagnosis of COVID-19 within the last 28 days (antigen test or RT-PCR). In this situation, vaccination can be postponed until the participant completes 30 days;
* Report of fever within 72 hours prior to vaccination (inclusion can be postponed until the participant completes 72 hours without fever and COVID-19 is discarded);
* Having received live attenuated virus vaccine in the last 28 days or inactivated vaccine in the last 14 days prior to inclusion in the study;
* Any other condition that, in the opinion of the Principal Investigator or its medical representative, could jeopardize the safety or rights of a potential participant or prevent them from complying with this protocol;
* Pregnancy or lactation.

Type of study/study design: Experimental, single-arm study in participants with comorbidities, previously immunized with 2 doses of CoronaVac, who will receive a booster vaccine with 1 dose of the Oxford/AstraZeneca vaccine.

Sample size: all active participants from the COVACManaus study (up to 5071)

Primary outcome: Detection and titration of antibodies against SARS-CoV-2 before (D0), at D90 and D180 after booster vaccination

Secondary outcomes:

* Profile of the cell-mediated immune response in a subgroup of participants, before (D0), at D90 and D180 after booster vaccination;
* Ability to neutralize antibodies in a subgroup of participants before (D0), in D90 and D180 after the vaccine booster;
* Memory cell populations in a subgroup of participants before (D0), in D90 and D180 after booster vaccination.
* Detection and titration of antibodies against SARS-CoV-2 and its association with the history of physical activity or sedentary lifestyle.

ELIGIBILITY:
Inclusion criteria:

* Have voluntarily participated and be in regular follow-up monitoring by the COVACMANAUS study;
* Have completed the vaccination schedule with 2 doses of CoronaVac, as per the COVACMANAUS study protocol for at least 180 days (+/- 30 days);
* Demonstrate availability to be followed during the follow-up period defined in the study, through visits, telephone contacts or other digital means of communication;
* Accept to participate in this new study for 6 (six) months.

Exclusion criteria

* Confirmed diagnosis of COVID-19 within the last 28 days (antigen test or RT-PCR). In this situation, vaccination can be postponed until the participant completes 30 days;
* Report of fever within 72 hours prior to vaccination (inclusion can be postponed until the participant completes 72 hours without fever and COVID-19 is discarded);
* Having received live attenuated virus vaccine in the last 28 days or inactivated vaccine in the last 14 days prior to inclusion in the study;
* Any other condition that, in the opinion of the Principal Investigator or its medical representative, could jeopardize the safety or rights of a potential participant or prevent them from complying with this protocol;
* Pregnancy or lactation.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4446 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Antibodies (detection and titration) against SARS-CoV-2 through quantitative test for total antibodies against viral nucleocapsid and IgG antibodies against Spike protein | change from baseline (Day 0) antibodies against SARS-CoV-2 at Day 90 (D90) and Day 180 (D180) after booster vaccination
  Detection and titration of antibodies against SARS-CoV-2 at baseline (Day 0) and at Day 90 and Day 180 after booster vaccination

SECONDARY OUTCOMES:
Profile of the cell-mediated immune response in a subgroup of participants through cell immunophenotyping, using the Flow Cytometry (FC) technique. | change from baseline profile (Day 0) of the cell-mediated immune response compared to Day 90 (D90) and Day 180 (D180) after booster vaccination
  • Profile of the cell-mediated immune response in a subgroup of participants, before (D0), at D90 and D180 after booster vaccination through cell immunophenotyping, using the Flow Cytometry (FC) technique. Memory T and B cell subpopulations will be labeled with monoclonal antibodies conjugated to pre-especified fluorochromes that bind to specific surface markers (clusters of differentiation) present in the populations of interest.
Ability of the serum from a subgroup of participants to neutralize antibodies though viral neutralization assay at baseline (Day 0) and at Day 90 and D180 after vaccine booster dose | change from baseline (Day 0) profile of the ability to neutralize antibodies in a subgroup of participants at Day 90 (D90) and Day 180 (D180) after booster vaccination
  • Ability to neutralize antibodies in a subgroup of participants, through the Viral Neutralization Test (VNT) consisting of cultured Vero CCL-81 cells, inactivated serial diluted serum and fixation.
Quantification of memory cell populations in a subgroup of participants | change from baseline (Day 0) memory cell populations in a subgroup of participants at Day 90 (D90) and Day 180 (D180) after booster vaccination
  • Profile of memory populations by cellular immunophenotyping in a subgroup of participants at baseline (Day 0) and in Day 90 and Day 180 after booster vaccination.
Physical activity and its relationship with the acquisition of antibodies against SARS-CoV-2 after booster vaccination against SARS-CoV-2. | change from baseline (Day 0) antibodies against SARS-CoV-2 at Day 90 (D90) and Day 180 (D180) after booster vaccination and it relationship with the history of physical activity
  • Detection and titration of antibodies against SARS-CoV-2 and relationship with the history of physical activity during the follow-up period. To access physical activity the International Physical Activity Questionnaire (IPAQ) will be used and combined with the Duke Activity Status Index (DASI) questionnaire for sedentary lifestyle.
Sedentary lifestyle and its relationship with the acquisition of antibodies against SARS-CoV-2 after booster vaccination against SARS-CoV-2. | change from baseline (Day 0) antibodies against SARS-CoV-2 at Day 90 (D90) and Day 180 (D180) after booster vaccination and it relationship with the history of sedentary lifestyle
  • Detection and titration of antibodies against SARS-CoV-2 and relationship with the history of sedentary lifestyle during the follow-up period. To access the sedentary lifestyle the Duke Activity Status Index (DASI) questionnaire will be used and combined with International Physical Activity Questionnaire (IPAQ) for physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Lacerda, PhD, Principal Investigator — Fundação de Medicina Tropical Dr. Heitor Vieira Dourado
Locations (1):
- Fundação de Medicina Tropical Dr Heitor Vieira Dourado, Manaus, Amazonas, Brazil